CLINICAL TRIAL: NCT04938882
Title: Effect of Ultrasound-guided Transversus Abdominis Plane Block With Compound Lidocaine on Postoperative Pain in Patients Undergoing Gynecological Laparotomy：a Randomized Double-blind Controlled Trial
Brief Title: Effect of Transversus Abdominis Plane Block With Compound Lidocaine on Pain After Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang013
Record Dates: First submitted 2021-06-22; First posted 2021-06-24 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Pain
Keywords: Compound lidocaine; Ropivacaine; pain intensity; Transversus abdominis plane block
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Saline Solution; Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal saline in transversus abdominis plane block (Placebo Comparator): Before the induction of anesthesia, normal saline is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Normal saline
- Ropivacaine in transversus abdominis plane block (Active Comparator): Before the induction of anesthesia, 0.375% ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Ropivacaine
- Compound lidocaine at low-concentration in transversus abdominis plane block (Active Comparator): Before the induction of anesthesia, 0.4% compound lidocaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Compound lidocaine at low concentration
- Compound lidocaine at high-concentration in transversus abdominis plane block (Active Comparator): Before the induction of anesthesia, 0.6% compound lidocaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Interventions: Drug: Compound lidocaine at high concentration

INTERVENTIONS:
Drug: Normal saline — Before the induction of anesthesia, normal saline is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: 0. 9% Sodium Chloride Injection
  Arms: Normal saline in transversus abdominis plane block
Drug: Ropivacaine — Before the induction of anesthesia, 0.375% ropivacaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: Ropivacaine Hydrochloride Injection
  Arms: Ropivacaine in transversus abdominis plane block
Drug: Compound lidocaine at low concentration — Before the induction of anesthesia, 0.4% compound lidocaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: Compound Hydrochloride Lidocaine Injection
  Arms: Compound lidocaine at low-concentration in transversus abdominis plane block
Drug: Compound lidocaine at high concentration — Before the induction of anesthesia, 0.6% compound lidocaine is used for bilateral transversus abdominis plane block in a volume of 20 mL of each side
  Other Names: Compound Hydrochloride Lidocaine Injection
  Arms: Compound lidocaine at high-concentration in transversus abdominis plane block

SUMMARY:
Purpose:

To explore effects of ultrasound-guided transversus abdominis plane block with compound lidocaine on postoperative pain after gynecological laparotomy.

DETAILED DESCRIPTION:
Poor post-surgical pain control is a leading factor that hinders the physical rehabilitation, and causes acute cognitive impairment and chronic pain syndrome. Recently, the multimodal analgesia strategies to minimise opioid-related side effects are highly desirable in open surgical procedures. The transversus abdominis plane block is a novel technique involving injection of local anaesthetic between the internal oblique and the transversus abdominis muscles of the abdominal wall. Although ropivacaine is most commonly used for this technique, the analgesic duration remains not dissatisfied. Compared with ropivacaine, compound lidocaine injection has a better and longer analgesic activity since it contains menthol and ethanol with appropriate concentrations. However, whether compound lidocaine injection is efficiency in the transversus abdominis plane block for abdominal open sugery lacks investigations. Herein, we will evaluate the efficacy of ultrasound-guided transversus abdominis plane (USG-TAP) block with compound lidocaine injection for postoperative analgesia in patients undergoing gynecological laparotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo gynecological laparotomy under general anesthesia
2. Subject's American Society of Anesthesiologists physical status is I-II.
3. The subject's parent/legally authorized guardian has given written informed consent to participate.

Exclusion Criteria:

1. Subject has a diagnosis of bronchial asthma, coronary heart disease, severe hypertension, renal failure or liver failure.
2. Subject has a diagnosis of Insulin dependent diabetes.
3. Subject is allergy and contraindication to local anesthetics or any components of local anesthetics.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre- existing therapy with opioids, intake of any analgesic drug within 48 hours before surgery.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Subject is pregnant or breast-feeding.
7. Subject is obese (body mass index >30kg/m^2).
8. Subject is incapacity to comprehend pain assessment and cognitive assessment.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Pain Score (NRS) | 72 hours after surgery
  The pain score at rest or after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.

SECONDARY OUTCOMES:
Time of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Total Dose of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of sufentanyl.
Cumulative Sufentanyl Consumption | 72 hours after surgery
  Each patient was administered analgesics using a PCA (Patient-controlled analgesia) pump containing sufentanil (200μg) in normal saline at a total volume of 200 ml after leaving PACU (Postanesthesia care unit). This device was set to deliver a basal infusion of 2 ml/h and bolus doses of 0.5 ml with a 15-min lockout period. Sufentanyl cumulative consumption is recorded 72 hours postoperatively
Occurrence of Side Effects | 72 hours after surgery
  Occurrence of side effects: nausea, vomiting, dizziness, headache, shivering, pruritus
Normalized Area of Hyperalgesia Around the Incision | 72 hours after surgery
  The skin around the incision is stimulated in steps of 5 mm at intervals of 1 s starting outside of the hyperalgesic area in the direction of the incision. The distance from the incision to the first point where a 'painful', 'sore' or 'sharper' feeling occurred is measured and noted. This measurement is repeated at predefined radial lines around the incision. To eliminate the variable length of incision, this length is subtracted from the longer diameter leaving four radial distances from the end and from the middle of the incision. The normalized area of hyperalgesia is calculated by summing up the areas of the remaining four triangles measured by and Von Frey filament.
The onset time of sensory block | 30 minutes after transversus abdominis plane block
  Sensory block was assessed using a cold test (2 = normal sensation, 1 = decreased cold sensation compared, 0 = loss of cold sensation) on the bilateral anterior abdomen between the median line and linea semiluminaris from T7-T12. The sensation was compared with the sensation to cold at ipsilateral lateral thoracic region of T4-T5.
Diffusion area of local anesthetics after transversus abdominis plane block | 30 minutes after transversus abdominis plane block
  Diffusion area of local anesthetics after transversus abdominis plane block was calculated under ultrasound assistance .
Apfel score | The day before the surgery
  The Apfel score was recorded for evaluating risk for developing postoperative nausea and vomiting (PONV).
Mean time until passage of flatus | 72 hours after surgery
  Gastrointestinal motility was evaluated by recording mean time until passage of flatus

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran DQ, Bravo D, Leurcharusmee P, Neal JM. Transversus Abdominis Plane Block: A Narrative Review. Anesthesiology. 2019 Nov;131(5):1166-1190. doi: 10.1097/ALN.0000000000002842. PMID 31283738
- [Background] Ma N, Duncan JK, Scarfe AJ, Schuhmann S, Cameron AL. Clinical safety and effectiveness of transversus abdominis plane (TAP) block in post-operative analgesia: a systematic review and meta-analysis. J Anesth. 2017 Jun;31(3):432-452. doi: 10.1007/s00540-017-2323-5. Epub 2017 Mar 7. PMID 28271227
- [Derived] Zhang L, Jia Z, Gao T, Wang Y, Zhao Y, Li J, Yu Y, Li Q, Wang G. A randomized controlled trial evaluating the effects of transversus abdominis plane block with compound lidocaine hydrochloride injection on postoperative pain and opioid consumption and gastrointestinal motility in patients undergoing gynecological laparotomy. Front Mol Neurosci. 2023 Jan 25;16:967917. doi: 10.3389/fnmol.2023.967917. eCollection 2023. PMID 36760605